CLINICAL TRIAL: NCT00239954
Title: Fixed Dose Comparison of Escitalopram Combination in Adult Patients With Major Depressive Disorder
Brief Title: Escitalopram Combination Comparison Study for Adult Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmacology Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRI#591 & #592
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of an escitalopram combination treatment compared to single treatments, and to placebo in patients with major depressive disorder.

DETAILED DESCRIPTION:
Both active drugs being tested, alone and in combination, in this study are currently available antidepressants. However, the doses used in this study are lower than the standard approved doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) diagnostic criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 12 weeks in duration.

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* Patients who currently meet DSM-IV criteria for : a. bipolar disorder; b. schizophrenia or any psychotic disorder; c. obsessive-compulsive disorder; d. mental retardation or any pervasive developmental disorder or cognitive disorder.
* Patients who are considered a suicide risk.
* Patients with a history of seizure disorder, or any history of seizure, stroke, significant head injury, or any other condition that predisposes toward risk of seizure.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-03

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD)

CONTACTS AND LOCATIONS:
Overall Officials: Jon F. Heiser, MD, Principal Investigator — Pharmacology Research Institute; Nader Oskooilar, MD, Principal Investigator — Pharmacology Research Institute
Locations (4):
- United States (4):
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pharmacology Research Institute, Northridge, California
  - Pharmacology Research Institute, Riverside, California